CLINICAL TRIAL: NCT04585971
Title: A Study on Hemodynamic Relationship Including Cerebral Blood Flow Using Phase Contrast and Signal Intensity Gradient of Brain Magnetic Resonance Imaging, and Carotid Doppler Ultrasound
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Chonbuk National University Hospital (Other)
Collaborators: Medi Image, Inc (Unknown)
Responsible Party: Principal Investigator, Chan-Hyuk Lee, Professor, Chonbuk National University Hospital
Other Study IDs: SIGBF
Record Dates: First submitted 2020-10-06; First posted 2020-10-14 (Actual); Last update posted 2020-10-14 (Actual); Status verified 2020-10

CONDITIONS: Cerebral Blood Flow
Keywords: Endothelial shear stress; signal-intensity gradient; phase contrast MRI; Time-of-Flight MRI; Carotid Doppler sonography

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Subjects: Cerebral blood flow of a subject is measured using three methods in both common carotid and vertebral arteries. 1) Phase-contrast MR 2) Doppler sonography 3) Signal Intensity Gradient (SIG) To determine whether there is a correlation between the measured values, the correlation coefficient is calculated and analyzed.
  Interventions: Diagnostic Test: Signal intensity gradient

INTERVENTIONS:
Diagnostic Test: Signal intensity gradient — Signal intensity gradient:
  In time-of-flight (TOF) MRA, The signal intensities at the iso-point (Φa; signal intensity at position A [Xa] along the arterial contour line) and at the inner point (Φb; signal intensity at position B [Xb]) were calculated by using a trilinear interpolation algorithm based on the positions and signal intensities in the eight neighboring voxels. The signal intensities of TOF-MRA were normalized to eliminate the offset and scale effects across the MRA datasets of participants. For each iso-point (position A), the SIG was calculated from the difference in signal intensities between points A and B as follows:
  Scalar SIG, SI/mm = (Φb - Φa) / │Xb - Xa│ (1)
  Vector SIG, SI/mm = (Φb - Φa) n / │Xb - Xa│ (2)
  Other Names: Time-of-flight magnetic resonance imaging; Carotid Doppler sonography

SUMMARY:
Cerebral blood flow measurement, which is applied to patients with cerebrovascular-related diseases, provides useful information about hemodynamic status. There was a method using Doppler ultrasound and phase contrast (PC) MRI, but it was not widely used in clinical practice due to limitations in reproducibility between examiners, complexity of procedure, and time-intensive protocol. We intend to measure cerebral blood flow through the signal-intensity gradient (SIG) technique using Time-of-Flight (TOF) of brain magnetic resonance imaging, which can compensate for the shortcomings of the existing research methods. In addition, by analyzing the correlation with the previous methods, Doppler ultrasound and PC MRI, we will evaluate the effectiveness of our new method.

ELIGIBILITY:
Inclusion Criteria:

1. Patients 18 years of age or older who have been admitted to the neurology department due to a stroke, and those who have already performed brain magnetic resonance imaging
2. Among the patients (1) who underwent carotid artery Doppler ultrasound
3. Patients who fully understand the research objectives and procedures and wish to participate in clinical research voluntarily
4. If a patient is not fully understood due to a decrease in awareness or consciousness, the consent of the legal representative is required

Exclusion Criteria:

1. Patients whose extracranial artery occlusion or severe stenosis was confirmed in brain magnetic resonance images.
2. Those who judge that the subject is unsuitable for participation in clinical research due to other reasons.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted to the neurology department of a tertiary center
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2020-09-03 (Actual); Primary Completion 2021-01-31 (Estimated); Study Completion 2021-01-31 (Estimated)

PRIMARY OUTCOMES:
Cerebral blood flow correlation | After completion of recruitment, average 1 year
  Cerebral blood flow correlation between 3 tests (SIG, PC MR, US)

CONTACTS AND LOCATIONS:
Overall Officials: Chan-Hyuk Lee, Prof., Principal Investigator — Jeonbuk National University Hospital
Locations (1):
- Jeonbuk National University Hospital, Jeonju, Jeollabuk-do, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Han KS, Lee SH, Ryu HU, Park SH, Chung GH, Cho YI, Jeong SK. Direct Assessment of Wall Shear Stress by Signal Intensity Gradient from Time-of-Flight Magnetic Resonance Angiography. Biomed Res Int. 2017;2017:7087086. doi: 10.1155/2017/7087086. Epub 2017 Aug 16. PMID 28900625
- [Background] Lee WJ, Jeong SK, Han KS, Lee SH, Ryu YJ, Sohn CH, Jung KH. Impact of Endothelial Shear Stress on the Bilateral Progression of Unilateral Moyamoya Disease. Stroke. 2020 Mar;51(3):775-783. doi: 10.1161/STROKEAHA.119.028117. Epub 2019 Dec 20. PMID 31856692
- [Background] Jeong SK, Lee JY, Rosenson RS. Association between Ischemic Stroke and Vascular Shear Stress in the Carotid Artery. J Clin Neurol. 2014 Apr;10(2):133-9. doi: 10.3988/jcn.2014.10.2.133. Epub 2014 Apr 23. PMID 24829599
- [Derived] Lee CH, Lee SH, Kwak HS, Rosenson RS, Jeong SK, Jung KH. Arterial flow volume measurement using signal intensity gradient versus phase contrast. Sci Rep. 2025 Dec 29;15(1):44848. doi: 10.1038/s41598-025-28379-7. PMID 41461703
- [Derived] Lee CH, Lee SH, Kwak HS, Kwak YG, Rosenson RS, Cho YI, Jeong SK. Validation of Signal Intensity Gradient from TOF-MRA for Wall Shear Stress by Phase-Contrast MR. J Imaging Inform Med. 2024 Jun;37(3):1248-1258. doi: 10.1007/s10278-024-00991-5. Epub 2024 Feb 8. PMID 38332403